CLINICAL TRIAL: NCT00438048
Title: Xerostomy Treatment in Patients With Sjogren's Syndrome in Chile :A Double Blind Control Trial Comparing Orally Pilocarpine Drops and Artificial Saliva
Brief Title: A Comparison of Orally Pilocarpine and Artificial Saliva in Xerostomy Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Formulario MAgistral Farmacias Ahumada (Unknown)
Responsible Party: Cristian Vera Kellet, Pontificia Universidad Católica de Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAVK-130108245-1
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Primary Sjogren; Secondary Sjogren; Xerostomia
Keywords: Pilocarpine; Artificial saliva; Xerostomia; Xerostomy; Primary Sjogren; Secondary Sjogren
MeSH Terms: conditions — Xerostomia | interventions — Pilocarpine; Saliva, Artificial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- a,b (Active Comparator): Compare Pilocarpine and Artificial saliva
  Interventions: Procedure: pilocarpine; Drug: Artificial Saliva

INTERVENTIONS:
Procedure: pilocarpine — or secondary symptomatic SS with clinically significant dry mouth were randomized to receive either 5 mg oral Pilocarpine solution (5ml) or artificial saliva (5 ml) 3 times a day for 12 weeks
  Other Names: Artificial saliva
Drug: Artificial Saliva — 5ml 3 times daily
  Other Names: pilocarpine

SUMMARY:
The purpose of this study is to assess and compare the safetyness and efficacy of pilocarpine drops versus artificial saliva as symptomatic treatment for dry mouth and dry eyes caused by SS in a multicenter, doubleblind, controlled trial.

DETAILED DESCRIPTION:
Title:

Xerostomy treatment in patients with Sjogren's syndrome in Chile :A double blind control trial comparing orally Pilocarpine drops and Artificial Saliva

Authors:

Cristian Vera Kellet, Mirtha Cifuentes Mutinelli. Affiliations: Pontificia Universidad Catolica de Chile

BACKGROUND Sjogren's syndrome (SS) is characterized by diminished exocrine secretions with the resultant xerostomia and xerophthalmia due to slowly progressive infiltration of lacrimal and salivary glands by inflamatory cells.

OBJECTIVE: To assess and compare the safetyness and efficacy of pilocarpine drops versus artificial saliva as symptomatic treatment for dry mouth and dry eyes caused by SS in a multicenter, doubleblind, controlled trial.

SUBJECTS AND METHODS After providing written informed consent, 72 patients with primary or secondary SS and clinically significant dry mouth and dry eyes will be randomized to receive either 5-mg pilocarpine drops, or artificial saliva 3 times daily for 12 weeks. Global evaluation and subjective responses of patients will be assessed by questionnaires with visual analog scales or categorical checkboxes. All patients will be submited to anxiety and psicological test before and after 12 weeks. Whole-mouth salivary flow and lacrimal flow will be measured using Schirmer test.

ELIGIBILITY:
Inclusion Criteria:

* Patiens over 18 years, with primary or secondary Sjogren's Syndrome and xerostomia.

Exclusion Criteria:

* Patiens with cardiac, pulmonary, renal, gastric diseases,
* Patients with diabetes, glaucoma, Multipleesclerosis,
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2006-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To assess and compare the safetyness and efficacy of pilocarpine drops versus artificial saliva as symptomatic treatment for dry mouth and dry eyes caused by SS in a multicenter, doubleblind, controlled trial. | 12 weeks

SECONDARY OUTCOMES:
Determine on a subjetive manner wich treatment is better fot patients. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Vera-Kellet, MD, Principal Investigator — UDA Dermatologia, Escuela de Medicina, Pontificia Universidad Catolica de Chile
Locations (1):
- Unidad Docente Asociada Dermatologia. Escuela de MEdicina Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Papas AS, Sherrer YS, Charney M, Golden HE, Medsger TA Jr, Walsh BT, Trivedi M, Goldlust B, Gallagher SC. Successful Treatment of Dry Mouth and Dry Eye Symptoms in Sjogren's Syndrome Patients With Oral Pilocarpine: A Randomized, Placebo-Controlled, Dose-Adjustment Study. J Clin Rheumatol. 2004 Aug;10(4):169-77. doi: 10.1097/01.rhu.0000135553.08057.21. PMID 17043506
- [Background] Al-Hashimi I. Xerostomia secondary to Sjogren's syndrome in the elderly: recognition and management. Drugs Aging. 2005;22(11):887-99. doi: 10.2165/00002512-200522110-00001. PMID 16323968
- [Background] Masters KJ. Pilocarpine treatment of xerostomia induced by psychoactive medications. Am J Psychiatry. 2005 May;162(5):1023. doi: 10.1176/appi.ajp.162.5.1023. No abstract available. PMID 15863819
- [Background] Gotrick B, Akerman S, Ericson D, Torstenson R, Tobin G. Oral pilocarpine for treatment of opioid-induced oral dryness in healthy adults. J Dent Res. 2004 May;83(5):393-7. doi: 10.1177/154405910408300508. PMID 15111631
- [Background] Hendrickson RG, Morocco AP, Greenberg MI. Pilocarpine toxicity and the treatment of xerostomia. J Emerg Med. 2004 May;26(4):429-32. doi: 10.1016/j.jemermed.2003.09.013. PMID 15093850
- [Background] Solans R, Bosch JA, Selva A, Simeon CP, Fonollosa V, Vilardell M. [Usefulness of oral pilocarpin therapy in the treatment of xerostomia and xerophthalmia in patients with primary Sjogren's syndrome]. Med Clin (Barc). 2004 Feb 28;122(7):253-5. doi: 10.1016/s0025-7753(04)75314-2. Spanish. PMID 15012873
- [Background] Tsifetaki N, Kitsos G, Paschides CA, Alamanos Y, Eftaxias V, Voulgari PV, Psilas K, Drosos AA. Oral pilocarpine for the treatment of ocular symptoms in patients with Sjogren's syndrome: a randomised 12 week controlled study. Ann Rheum Dis. 2003 Dec;62(12):1204-7. doi: 10.1136/ard.2002.003889. PMID 14644860
- [Result] Wu CH, Hsieh SC, Lee KL, Li KJ, Lu MC, Yu CL. Pilocarpine hydrochloride for the treatment of xerostomia in patients with Sjogren's syndrome in Taiwan--a double-blind, placebo-controlled trial. J Formos Med Assoc. 2006 Oct;105(10):796-803. doi: 10.1016/S0929-6646(09)60266-7. PMID 17000452
- [Result] Brito-Zeron P, Ramos-Casals M, Nardi N, Font J. [Results of the treatment with oral pilocarpine in 100 patients with primary Sjogrens syndrome]. Med Clin (Barc). 2006 Apr 29;126(16):637. doi: 10.1157/13087738. No abstract available. Spanish. PMID 16759558
- [Result] Aframian DJ, Helcer M, Livni D, Markitziu A. Pilocarpine for the treatment of salivary glands' impairment caused by radioiodine therapy for thyroid cancer. Oral Dis. 2006 May;12(3):297-300. doi: 10.1111/j.1601-0825.2005.01195.x. PMID 16700739
- [Result] Aragona P, Di Pietro R, Spinella R, Mobrici M. Conjunctival epithelium improvement after systemic pilocarpine in patients with Sjogren's syndrome. Br J Ophthalmol. 2006 Feb;90(2):166-70. doi: 10.1136/bjo.2005.078865. PMID 16424527